CLINICAL TRIAL: NCT05512637
Title: Screening for Neurodevelopmental Disorders in Siblings of Children With Autism Diagnosed in Tertiary Centers
Acronym: FRATSA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Principal Investigator, Véronique GONNIER, child psychiatrist, University Hospital, Montpellier
Other Study IDs: RECHMPL21_0358
Record Dates: First submitted 2022-07-26; First posted 2022-08-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Siblings; Neurodevelopmental Disorders
Keywords: Siblings; Screening; Autism Spectrum Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- neurodevelopmental disorders: Step 1 - Screening: the targeted sample is the siblings of the autistic children, these siblings being at risk of neurodevelopmental disorders.
  Step 2 - Clinical interview: All the children with a positive screening.
  Interventions: Diagnostic Test: Step 1 - Screening ; Step 2 - Clinical interview

INTERVENTIONS:
Diagnostic Test: Step 1 - Screening ; Step 2 - Clinical interview — Step 1: screening is performed by online parental questionnaires (SRS-2, Identidys scale, DCDQ, parental concerns questionnaire ) via a web platform. Parents and registered doctors will be informed by mail in case of negative screening; In case of positive screening, they will be called by phone in order to give them the results and to invite them for a clinical and semi-structured interview.
  Step 2: The semi-structured interview will be performed by a psychologist specialized in NDD in order to clinically confirm the results of the screening and refer the child to care and interventions, by mail to the registered doctor. Around 12 months after this interview, parents will be called by phone to collect a description of the referral and their satisfaction about the screening process.

SUMMARY:
In this study, a selective and multi-stages screening for neurodevelopmental disorders (NDD) in siblings of children with a confirmed ASD is done. The main aims are to estimate the prevalence of NDD among siblings and to evaluate the feasibility and acceptability of a standardized screening procedure.

DETAILED DESCRIPTION:
Although NDD are frequent among siblings of children with ASD, their developmental screening is not yet sufficiently organized in routine practice. The needs and the characteristics of these siblings have yet to be better understood in order to define their developmental surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Step 1: Brothers or sisters (including stepsisters and brothers); aged between 2 and 16 years; living in Occitanie; informed and express consent of parents ; affiliated to social security.
* Step 2: step 1 positive screening or parental concerns for child's development ; parental signed informed consent.

Exclusion Criteria:

* Parents (or child) refusal to participate; adopted brother or sister. Do not speak French

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The expected number of children is 384 children (142 with NDD and 242 without NDD).
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of family participation | 12 months
  Families' participation rate and, among participants, number of children with a NDD diagnosis at the end of the screening study.

SECONDARY OUTCOMES:
Sensibility, specificity, positive predictive values (PPV) and negative predictive values (NPV) of the screening procedure | 12 months
Percentage of satisfied parents | 12 months
  Estimate the level of satisfaction of parents who participated in the screening with the parental satisfaction score via the Visual Analog Scale (VAS).
  VAS is a scale from 0 (not at all satisfied) to 100 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique GONNIER, Dr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baghdadli A, Audras-Torrent L, Rattaz C, Gonnier V, Ferrando L, Michelon C, Odoyer R, Maffre T, Picot MC. Multistage screening process for neurodevelopmental disorders in siblings of children with autism: the FRATSA protocol study. BMJ Open. 2023 Jan 30;13(1):e066520. doi: 10.1136/bmjopen-2022-066520. PMID 36717133
- Available data/document: Study Protocol — https://bmjopen.bmj.com/content/14/11/e084110